CLINICAL TRIAL: NCT06163014
Title: My Symptoms: a Before-After Evaluation of an eHealth and GP Assisted Programme for Persistent Symptoms in Primary Care (eASY)
Brief Title: My Symptoms: an eHealth and GP Assisted Programme for Persistent Symptoms in Primary Care
Acronym: eASY
Status: Recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Rosendal, Principal Investigator, senior researcher, MD, PhD, Aarhus University Hospital
Other Study IDs: 1-10-72-222-22
Record Dates: First submitted 2023-06-08; First posted 2023-12-08 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Persistent Physical Symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with persistent physical symptoms consulting their GP and referred to the My Symptoms eHealth programme.
  Interventions: Behavioral: My Symptoms eHealth programme

INTERVENTIONS:
Behavioral: My Symptoms eHealth programme — My Symptoms supports patients' self-efficacy and behavioural changes. The programme is activated by the patient after prescription by the GP. The patient is free to choose relevant tasks corresponding to wishes, needs/requirements and own perspectives.
  Summary of content:
  1. Symptom explanations and facts about frequent symptoms including brief animated explanations
  2. Physical energy (sleep, diet and activity)
  3. Working with resources and strain in everyday life
  4. Values and choices (meaning and existential issues)
  5. Thoughts
  6. Feelings (emotion regulation)
  7. Self-care (attention incl. mindfulness and audio exercises)
  8. Preparation for a follow-up visit with the GP and relapse prevention. The above modules connect to four general tools: symptom registration, 'don't break the chain', goal setting staircase and notebook.
  After 6 weeks: Voluntary GP follow-up consultation. After 8 weeks: End-of-treatment.

SUMMARY:
The project 'My Symptoms' is part of a large research programme: eHealth and GP-assisted self-help interventions for persistent physical symptoms (eASY). See www.mine-symptomer.dk.

The research programme is an ambitious and dedicated effort aiming at improvement of functioning and quality of life for individuals with persistent physical symptoms (PPS) and prevention of the development of chronic functional disorders and associated loss of working capacity and high use of health care. At present, access to specialized treatment of PPS is very limited and treatment capacity in general practice is restricted to brief consultations - often with poor opportunity to make a treatment plan for symptoms. As part of the research programme, the investigators have developed a web-based self-help programme for patient with PPS. This treatment programme is prescribed by the patient's general practitioner (GP). Only GPs who have participated in a short introduction course will be allowed for prescriptions.

The investigators have applied a high degree of user involvement (GPs and patients) in the development process but there is a need to evaluate how the new treatment programme is in fact adopted by GPs and patients.

With this study, the investigators wish to follow the national implementation using a before-after study design describing uptake and effects on GPs, patients and the health care system.

DETAILED DESCRIPTION:
The project aims to evaluate the uptake and effects of the new self-help programme for PPS, the My Symptoms programme, prescribed and followed up by GPs.

Specific objectives are to:

1. Describe the use of the programme during routine care. This includes

   1. Determination of the number of patients per GP who access the programme after prescription from their GPs (adoption)
   2. A description of how often the follow-up consultation is completed according to the patients.
2. Explore patient characteristics (appropriateness)
3. Describe patients' engagement with the programme with regard to time and frequency of access to modules and tools (fidelity)
4. Evaluate effects on patients' health, quality of life, functioning and satisfaction with care
5. Estimate effects on patients' use of health care services
6. Estimate effects on patients' work productivity
7. Estimate possible effects on health care costs provided the intervention is fully disseminated nationally.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 (target population for the programme)
* The consultation targets symptom complaints
* Listed with participating practice.

Exclusion Criteria:

* Symptoms are acute (not persistent) and there is no need for this intervention
* Symptoms must primarily be treated by medicine or surgery
* Patient severely affected by other disease
* Not eligible due to language or cognitive problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only patients who consult their GP will be eligible for participation. Patients will need a referral from their GP to be able to access the 'My Symptoms' programme using a specific code. All patients who consent to participate and login to the programme will be included in the present study. The GP will assess whether prescription of the 'My Symptoms' programme is relevant. As a guide for this assessment, the GP will be provided with the inclusion and exclusion criteria during their training programme.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in symptom intensity | Baseline to end of treatment (week 8)
  Symptom intensity measured by a numeric rating scale (0-10)
Change in symptom interference | Baseline to end of treatment (week 8)
  Symptom interference measured by a numeric rating scale (0-10)

SECONDARY OUTCOMES:
Change in symptom intensity | Baseline to 3 months after end of treatment
  Symptom intensity measured by a numeric rating scale (0-10)
Change in symptom interference | Baseline to 3 months after end of treatment
  Symptom interference measured by a numeric rating scale (0-10)
Change in symptom burden | Baseline to end of treatment (week 8)
  Bodily Distress Syndrome (BDS) Checklist measuring symptom burden (0-100)
Change in symptom burden | Baseline to 3 months after end of treatment
  Bodily Distress Syndrome (BDS) Checklist measuring symptom burden (0-100)
Bodily Distress Syndrome | Baseline
  Bodily Distress Syndrome (BDS) Checklist measuring BDS (0/1)
Bodily Distress Syndrome | End of treatment (week 8)
  Bodily Distress Syndrome (BDS) Checklist measuring BDS (0/1)
Bodily Distress Syndrome | 3 months after end of treatment
  Bodily Distress Syndrome (BDS) Checklist measuring BDS (0/1)
Change in illness perception | Baseline to end of treatment (week 8)
  Brief Illness Perception Questionnaire (B-IPQ). Sum score (min 0; max 70). Lower scores indicate more positive illness perceptions.
Change in illness perception | Baseline to 3 months after end of treatment
  Brief Illness Perception Questionnaire (B-IPQ). Sum score (min 0; max 70). Lower scores indicate more positive illness perceptions.
Change in illness worry | Baseline to end of treatment (week 8)
  The revised version of the six-item Whiteley Index (WI-6-R). Sum score (min 0; max 24). Higher scores indicate higher illness worry.
Change in illness worry | Baseline to 3 months after end of treatment
  The revised version of the six-item Whiteley Index (WI-6-R). Sum score (min 0; max 24). Higher scores indicate higher illness worry.
Anxiety | Baseline
  Symptom Checklist Anxiety (SCL-ANX4). Sum score (min 0; max 16). Higher scores indicate higher impairment.
Anxiety | End of treatment (week 8)
  Symptom Checklist Anxiety (SCL-ANX4). Sum score (min 0; max 16). Higher scores indicate higher impairment by anxiety.
Anxiety | 3 months after end of treatment
  Symptom Checklist Anxiety (SCL-ANX4). Sum score (min 0; max 16). Higher scores indicate higher impairment by anxiety.
Depression | Baseline
  Symptom Checklist Depression (SCL-DEP6). Sum score (min 0; max 24). Higher scores indicate higher impairment by depression.
Depression | End of treatment (week 8)
  Symptom Checklist Depression (SCL-DEP6). Sum score (min 0; max 24). Higher scores indicate higher impairment by depression.
Depression | 3 months after end of treatment
  Symptom Checklist Depression (SCL-DEP6). Sum score (min 0; max 24). Higher scores indicate higher impairment by depression.
Distress | Baseline
  Symptom Checklist Distress (SCL-Distress8). Sum score (min 0; max 32). Higher scores indicate higher impairment by distress.
Distress | End of treatment (week 8)
  Symptom Checklist Distress (SCL-Distress8). Sum score (min 0; max 32). Higher scores indicate higher impairment by distress.
Distress | 3 months after end of treatment
  Symptom Checklist Distress (SCL-Distress8). Sum score (min 0; max 32). Higher scores indicate higher impairment by distress.
Change of hope | Baseline to end of treatment (week 8)
  One item from the Symptom Checklist (SCL)-90. Response categories ranging from 'not at all' (0) to 'very much' (4) (min 0; max 4). Higher scores indicate higher impairment by hopelessness.
Change of hope | Baseline to 3 months after end of treatment
  One item from the Symptom Checklist (SCL)-90. Response categories ranging from 'not at all' (0) to 'very much' (4) (min 0; max 4). Higher scores indicate higher impairment by hopelessness.
Change in stress | Baseline to end of treatment (week 8)
  Perceived Stress Scale 10-item version (PSS-10). Sum score (min 0; max 40). Higher scores indicate higher stress levels.
Change in stress | Baseline to 3 months after end of treatment
  Perceived Stress Scale 10-item version (PSS-10). Sum score (min 0; max 40). Higher scores indicate higher stress levels.
Change in limiting behaviour | Baseline to end of treatment (week 8)
  Behaviour Related to Illness Questionnaire (BRIQ), subscale. Sum score (min 0; max 24). Lower scores indicate a more adaptive symptom behaviour.
Change in limiting behaviour | Baseline to 3 months after end of treatment
  Behaviour Related to Illness Questionnaire (BRIQ), subscale. Sum score (min 0; max 24). Lower scores indicate a more adaptive symptom behaviour.
Change in all or nothing behaviour | Baseline to end of treatment (week 8)
  Behaviour Related to Illness Questionnaire (BRIQ), subscale. Sum score (min 0; max 28). Lower scores indicate a more adaptive symptom behaviour.
Change in all or nothing behaviour | Baseline to 3 months after end of treatment
  Behaviour Related to Illness Questionnaire (BRIQ), subscale. Sum score (min 0; max 28). Lower scores indicate a more adaptive symptom behaviour.
Change in confidence in performing activities in the context of PPS | Baseline to end of treatment (week 8)
  Adapted version of the Pain Self-Efficacy Questionnaire (PSEQ). Sum score (min 0; max 60). Higher scores indicate better self-efficacy.
Change in confidence in performing activities in the context of PPS | Baseline to 3 months after end of treatment
  Adapted version of the Pain Self-Efficacy Questionnaire (PSEQ). Sum score (min 0; max 60). Higher scores indicate better self-efficacy.
Change in health-related quality of life | Baseline to end of treatment (week 8)
  36-Item Short Form Health Survey (SF-36) (subscales and the physical (PCS) and mental (MCS) component summary scores). PCS and MCS will be transformed into scales ranging from 0 to 100 by the following expression: (patient raw score-lowest possible score)/(highest possible score-lowest possible score)×100. Higher scores express better health.
Change in health-related quality of life | Baseline to 3 months after end of treatment
  36-Item Short Form Health Survey (SF-36) (subscales and the physical (PCS) and mental (MCS) component summary scores). PCS and MCS will be transformed into scales ranging from 0 to 100 by the following expression: (patient raw score-lowest possible score)/(highest possible score-lowest possible score)×100. Higher scores express better health.
Health-related quality of life | Baseline
  The EuroQoL 5-domain 5-level (EQ-5D-5L). EQ-5D-5L health states will be summarised by a single summary number (index value), which reflects how good or bad the health state is according to the preferences of the general population. Index values will be derived according to the EuroQol Research Foundation manual for EQ-5D-5L.
Health-related quality of life | End of treatment (week 8)
  The EuroQoL 5-domain 5-level (EQ-5D-5L). EQ-5D-5L health states will be summarised by a single summary number (index value), which reflects how good or bad the health state is according to the preferences of the general population. Index values will be derived according to the EuroQol Research Foundation manual for EQ-5D-5L.
Health-related quality of life | 3 months after end of treatment
  The EuroQoL 5-domain 5-level (EQ-5D-5L). EQ-5D-5L health states will be summarised by a single summary number (index value), which reflects how good or bad the health state is according to the preferences of the general population. Index values will be derived according to the EuroQol Research Foundation manual for EQ-5D-5L.
Credibility related to the eHealth programme | Baseline
  One item measuring credibility. A scale ranging from 'not meaningful at all' (1) to 'highly meaningful' (10) is provided.
Expectancy related to the eHealth programme | Baseline
  One item measuring expectancy. A scale ranging from 'not efficient at all' (1) to 'highly efficient' (10) is provided.
Evaluation of the referral consultation | Baseline
  Questionnaire comprising 6 items. The items are scored on a five-point Likert-type scale ranging from 'bad' (1) to 'excellent' (5).
Evaluation of the eHealth programme | End of treatment (week 8)
  Questionnaire comprising 12 items. The items are scored on a five-point Likert-type scale representing the extent to which the patient find the programme easy to use or has experienced benefit. The scale ranges from 'not at all' (0) to 'to a very great extent' (4).
Recommendation of the eHealth programme | End of treatment (week 8)
  One item. The patient is asked to indicate whether he or she would recommend the treatment programme to a friend with similar problems. A VAS scale (0 ('not at all') - 10 ('highly recommend') is provided.
Evaluation of the follow up consultation | End of treatment (week 8)
  One item measuring satisfaction. The item is scored on a five-point Likert-type scale ranging from 'bad' (1) to 'excellent' (5).
Self-rated global health change | End of treatment (week 8)
  Patient Global Impression of Change (PGIC) scale. One item scored on a five point Likert-type scale ranging from 'Much worse' (1) to 'Much better' health (5).
Self-rated global health change | 3 months after end of treatment
  Patient Global Impression of Change (PGIC) scale. One item scored on a five point Likert-type scale ranging from 'Much worse' (1) to 'Much better' health (5).
Adverse events | End of treatment (week 8)
  Dichotomous outcome measure (0/1). Defined as a 50% worsening of symptoms as measured by the numeric rating scale (NRS) for symptom intensity
Adverse events | 3 months after end of treatment
  Dichotomous outcome measure (0/1). Defined as a 50% worsening of symptoms as measured by the numeric rating scale (NRS) for symptom intensity
Quality-adjusted life year (QALY) | 6 months after end of treatment
  QALY is a single reported value based on the change in patient's health-related quality of life measured with the EuroQoL 5-domain 5-level (EQ-5D-5L) and valued using Danish QALY-weights.
Changes in health care use | 6 months before baseline compared to 6 months after end of treatment
  Estimation of effects on patients' changes in use of health care services using Danish registers from a before-vs-after approach
Changes in productivity costs | 6 months before baseline compared to 6 months after end of treatment
  Changes in productivity costs i.e., the change in lost production due to changes in sick leaves and absence from work

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- See also: Project website — https://www.mine-symptomer.dk/